CLINICAL TRIAL: NCT03932838
Title: Descriptive Study of Multiligamentary Reconstruction of the Knee: Clinical Results and Postoperative Laxity by Dynamic Radiography.
Brief Title: Descriptive Study of Multiligamentary Reconstruction of the Knee
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Nicolas Pujol, Principal Investigateur, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P17/12_ Reconstruction
Record Dates: First submitted 2019-04-12; First posted 2019-05-01 (Actual); Last update posted 2019-05-01 (Actual); Status verified 2019-04

CONDITIONS: Injury, Knee
MeSH Terms: conditions — Knee Injuries | interventions — X-Rays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- clinical and radiologic evaluation (Experimental): Follow up post surgery: clinical and radiologic evaluation
  Interventions: Other: Clinical and radiologic evaluation

INTERVENTIONS:
Other: Clinical and radiologic evaluation — Follow up post surgery: clinical and radiologic evaluation

SUMMARY:
Evaluation of clinical results and postoperative laxity after single-stage reconstruction of multiligamentous lesions of the knee. Comparison of two types of transplant: allograft versus autograft.

There is currently little data in the clinical outcome literature after allograft reconstruction. There is one study reporting postoperative laxity assessed by dynamic radiography in the four planes (anterior, posterior, varus, valgus). No study compares postoperative laxity after allograft versus autograft reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated for one-time allograft or autograft reconstruction of multiligamentous knee injury
* >18 years old

Exclusion Criteria:

* Neurological or vascular injury during trauma.
* Fracture of the femur or both bones of the leg.
* Ligamentous lesion on the contralateral knee.
* History of surgery on the affected knee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Joint mobility of both knees | 2 years
  Postoperative knee function assessed by clinical examination
Postoperative laxity in varus, valgus, anterior and posterior drawer | 2 years
  Postoperative knee function assessed by clinical examination
Postoperative knee function assessed by scores | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- CH de Versailles, Le Chesnay, France

IPD SHARING:
Plan to Share IPD: No